CLINICAL TRIAL: NCT00494780
Title: An Open-labeled, Randomized, Two-dose, Parallel Group Trial of Ofatumumab, a Fully Human Monoclonal Anti-CD20 Antibody, in Combination With CHOP, in Patients With Previously Untreated Follicular Lymphoma (FL).
Brief Title: Ofatumumab (Humax-CD20) With CHOP (Cyclophosphamide,Doxorubicin, Vincristine, Predisolone) in Follicular Lymphoma (FL) Patients
Acronym: MUNIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111775; Hx-CD20-409 (Other: Genmab); The MUNIN trial
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma, Follicular
Keywords: CHOP (cyclophosphamide,doxorubicin,vincristine,prednisolone); ofatumumab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ofatumumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator 1 (Active Comparator): Each patient will receive a total of 6 infusions with ofatumumab in combination with CHOP every 3 weeks. The first infusion will be 300mg followed by 5 infusions of 500mg
  Interventions: Drug: Ofatumumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone, Prednisone or equivalent
- Active Comparator 2 (Active Comparator): Each patient will receive a total of 6 infusions with ofatumumab in combination with CHOP every 3 weeks. The first infusion will be 300mg followed by 5 infusions of 1000mg
  Interventions: Drug: Ofatumumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone, Prednisone or equivalent

INTERVENTIONS:
Drug: Ofatumumab — ofatumumab 300mg, 500mg or 1000mg should be diluted into 1000mL pyrogen free saline and administered as an IV infusion.Duration of infusion will be approximately 4 hours.Infusions should be given every 3 weeks until a total of 6 infusions has been given
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 iv for 1 day, 24-48h post-ofatumumab infusion start
  Other Names: CHOP
Drug: Doxorubicin — Doxorubicin : 50mg/m2 iv for 1 day, 24-48h post-ofatumumumab infusion start
  Other Names: CHOP
Drug: Vincristine — Vincristine : 1.4mg/m2 iv for 1 day, 24-48h post-ofatumumab infusion start
  Other Names: CHOP
Drug: Prednisolone, Prednisone or equivalent — 100mg p.o daily for 5 days, 24-48h post-ofatumumab infusion start
  Other Names: CHOP

SUMMARY:
To investigate the efficacy in two dose regimens of ofatumumab in combination with CHOP (cyclophosphamide,doxorubicin, vincristine,prednisolone) in previously untreated patients with Follicular Lymphoma (FL)

ELIGIBILITY:
Inclusion Criteria:

* Patient with Follicular Lymphoma (FL)
* Confirmed diagnosis of Follicular lymphoma
* 18 years or above
* Verbal and written information about the study

Exclusion Criteria:

* No previous treatment for Follicular Lymphoma
* Clinical suspicion that the Follicular Lymphoma has transformed to aggressive lymphoma
* Several diseases such as malignancies etc.
* Screening laboratory values
* Current participation in any other interventional clinical study
* Breast feeding women or pregnant women
* Women of childbearing potential not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Background] Czuczman MS, Hess G, Gadeberg OV, Pedersen LM, Goldstein N, Gupta I, Jewell RC, Lin TS, Lisby S, Strange C, Windfeld K, Viardot A; 409 Study Investigators. Chemoimmunotherapy with ofatumumab in combination with CHOP in previously untreated follicular lymphoma. Br J Haematol. 2012 May;157(4):438-45. doi: 10.1111/j.1365-2141.2012.09086.x. Epub 2012 Mar 13. PMID 22409295

RESULTS

PARTICIPANT FLOW:
Groups:
- 500 mg Ofatumumab + CHOP: Ofatumumab was given on Day 1 and CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone) on Day 3 of each 21-day cycle, with 300 milligrams (mg) in Cycle 1 and 500 mg in Cycles 2 to 6. Participants were followed up for 15 weeks during the Treatment period; then every 3 months for 24 months in the Follow-up period; then every 6 months until Month 60 or withdrawal from the study.
- 1000 mg Ofatumumab + CHOP: Ofatumumab was given on Day 1 and CHOP on Day 3 of each 21-day cycle, with 300 mg in Cycle 1 and 1000 mg in Cycles 2 to 6. Participants were followed up for 15 weeks during the Treatment period; then every 3 months for 24 months in the Follow-up period; then every 6 months until Month 60 or withdrawal from the study.
Period: Overall Study
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Started | 29 | 30
Completed | 18 | 17
Not Completed | 11 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew before Dosed | 0 | 1
Not completed — Progression of Study Disease | 7 | 8
Not completed — New Treatment | 2 | 2
Not completed — Non-compliance | 1 | 0
Not completed — Residual Tumour Mass | 0 | 1
Not completed — Insurance Issues | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 500 mg Ofatumumab + CHOP: Ofatumumab was given on Day 1 and CHOP on Day 3 of each 21-day cycle, with 300 mg in Cycle 1 and 500 mg in Cycles 2 to 6. Participants were followed up for 15 weeks during the Treatment period; then every 3 months for 24 months in the Follow-up period; then every 6 months until Month 60 or withdrawal from the study.
- Total: Total of all reporting groups
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who were exposed to trial drug irrespective of their compliance to the planned course of treatment.
  One participant was enrolled and randomized to receive 1000 mg Ofatumumab + CHOP, but withdrew prior to initiation of therapy.
  Years | 54.1 (11.4) | 53.7 (9.14) | 53.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who were exposed to trial drug irrespective of their compliance to the planned course of treatment.
  One participant was enrolled and randomized to receive 1000 mg Ofatumumab + CHOP, but withdrew prior to initiation of therapy.
  Participants
    Female | 14 | 21 | 35
    Male | 15 | 8 | 23
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in the Full Analysis Set (FAS), comprised of all participants who were exposed to trial drug irrespective of their compliance to the planned course of treatment.
  One participant was enrolled and randomized to receive 1000 mg Ofatumumab + CHOP, but withdrew prior to initiation of therapy.
  participants
    White | 29 | 27 | 56
    Hispanic or Latino | 0 | 2 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Complete Remission (CR) at Visit 26
Description: Participants were evaluated for response by an Independent Endpoint Review Committee in accordance with the standardized response criteria for NHL. Participants with CR were defined as those with the complete disappearance of all detectable clinical and radiographic evidence of disease.
Time Frame: Maximum of 23 months after the start of treatment
Population: FAS
Measure: Number; unit: participants
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
participants | 6 | 9

2. Secondary Outcome: Median Percent Change From Visit 1 (Screening, Week -2) in Tumor Size at Visit 33 (24 Months After the Last Infusion of Ofatumumab)
Description: The tumor size for a participant was computed as the sum of product of diameters (SPD) for the indicator lesions. Reduction in tumor size was calculated as percent change from Visit 1 until Visit 33, separately by radiologist 1 and radiologist 2. Percent change from Visit 1 (Screening, Week -2) = (value at Visit 33 minus value at Visit 1 divided by value at Visit 1) * 100.
Time Frame: Maximum of 24 months after the last infusion of Ofatumumab (Visit 33; median of 33.8 months)
Population: FAS. Participants were withdrawn from the study between Visits 1 and 33.
Measure: Median (Full Range); unit: Percent change in tumor size
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 17 | 16
Percent change in tumor size
  Radiologist 1 | -100 [-100 to 17.00] | -100 [-100 to -80.00]
  Radiologist 2 | -100 [-100 to -25.00] | -100 [-100 to -79.00]

3. Secondary Outcome: Time to New Anti-follicular Lymphoma (FL) Therapy
Description: Time to new FL therapy is defined as the time from randomization until the time of first administration of the new FL therapy other than ofatumumab. Time to new FL therapy will be censored if participants are lost to follow-up. The censoring date in such cases will be the date of the last attended visit at which the endpoint was assessed.
Time Frame: Followed up to 5 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
months | 47.2 [30.4 to NA] — There were too few participants; therefore, the upper limit of the CI could not be estimated. | NA [32.2 to NA] — There were too few participants; therefore, the median and the upper limit of the CI could not be estimated.

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization until progression or death.
Time Frame: Followed up to 5 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
months | 27.6 [15.1 to 28.3] | NA [21.3 to NA] — There were too few events for the median and upper limit of the CI to be estimated.

5. Secondary Outcome: Duration of Response
Description: The duration of response is defined as the time from the initial response (the first visit at which response was observed) to progression or death.
Time Frame: Followed up to 5 years
Population: FAS. Only those participants with a response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 26 | 29
months | 21.0 [13.3 to 26.2] | 25.0 [13.7 to NA] — There were too few events for the upper limit of the CI to be estimated.

6. Secondary Outcome: Percent Change From Visit 1 (Screening) in Peripheral CD19+ and CD20+ Cell Counts at Visit 33 (24 Months After the Last Infusion of Ofatumumab)
Description: The peripheral blood for each participant was collected and analyzed for CD19+ and CD20+ cell counts. CD19+ and CD20+ are B-cell types which are used as an index of a participant's response to treatment.
Time Frame: Maximum of 24 months after the last infusion of Ofatumumab (Visit 33; median of 33.8 months)
Population: FAS. Only those participants who provided samples at Visit 33 were analyzed.
Measure: Median (Full Range); unit: Percent change in cell counts
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 17 | 16
Percent change in cell counts
  CD19+ | 154.1 [-95 to 748] | 307.9 [-51 to 1767]
  CD20+ | 154.1 [-95 to 520] | 307.9 [-51 to 1767]

7. Secondary Outcome: Number of Participants Who Experienced Any Adverse Event (AEs) From First Treatment to Visit 33 (24 Months After Last Infusion)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. A list of AEs experienced in the study with a frequency threshold of 5% can be found in the AE section.
Time Frame: Up to 22 months after study start
Population: FAS
Measure: Number; unit: participants
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
participants | 29 | 29

8. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibodies (HAHA) at Visits 1, 28, and 33
Description: HAHA are indicators of immunogenicity to ofatumumab. Blood samples were drawn from participants at Visits 1, 28, and 33 for analysis of HAHA.
Time Frame: Visits 1 (Screening), 28 (9 months after last dose), and 33 (24 months after last dose)
Population: FAS. Participants dropped out of the study as the study progressed.
Measure: Number; unit: participants
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
participants
  Visit 1, n=29, 29 | 0 | 0
  Visit 28, n=18, 21 | 0 | 0
  Visit 33, n=16, 16 | 0 | 0

9. Secondary Outcome: Median Percent Change From Visit 1 (Screening) in Serum Complement (CH50) Levels at Visit 22
Description: The peripheral blood for each participant was collected and analyzed for serum complement CH50 levels. Cluster of Differentiation index 50 (CD50) is a human gene which is used as an index of immune response. CD50Percent change from Visit 1 (Screening, Week -2) = (value at Visit 22 minus value at Visit 1 divided by value at Visit 1) * 100.
Time Frame: Visit 1 (Screening, Week -2) and Visit 22 (Week 15)
Population: FAS. Only those participants who remained in the study at Visit 22 were analyzed.
Measure: Median (Full Range); unit: Percent change in serum complement CH50
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 24 | 28
Percent change in serum complement CH50 | 42.0 [-36 to 450] | 23.2 [-55 to 620]

10. Primary Outcome: Number of Participants With the Indicated Overall Best Response (OBR) at Visit 26 (3 Months After the Last Infusion of Ofatumumab)
Description: Based on standardized response criteria for NHL, responders included participants with CR (complete disappearance of all detectable clinical and radiographic evidence of disease), CRu (more than a 75% decrease in LN size compared to baseline), and PR (>=50% decrease in LN size and evidence of new lesions). Non-responders included participants with stable disease (SD; <50% decrease in LN size from baseline) and progressive disease (PD; >=50% increase in LN size and evidence of new lesions).
Time Frame: Maximum of 23 months after the start of treatment
Population: FAS
Measure: Number; unit: participants
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 29 | 29
participants
  Responder, CR | 6 | 9
  Responder, CRu | 10 | 7
  Responder, PR | 10 | 13
  Non-Responder, SD | 2 | 0
  Non-Responder, PD | 1 | 0

11. Secondary Outcome: Number of Participants Who Had a Conversion of BCL-2 t(14;18)-Positive to Negative by Polymerase Chain Reaction (PCR) in Peripheral Blood and Bone Marrow Aspirate and Its Durability Post-therapy
Description: This is a genetic prognostic marker of FL response. The former sponsor decided to not analyze these samples; therefore, no results are presented.
Time Frame: Maximum of 6 years follow-up
Population: FAS
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Cmax and Ctrough at the Sixth Infusion (Week 15, Visit 22)
Description: Cmax is defined as the maximum concentration of drug in plasma samples. Ctrough is defined as the trough plasma concentration (measured concentration at the end of a dosing interval [taken directly before next administration]).
Time Frame: Week 15 (Visit 22)
Population: FAS. Data were provided for the number of participants who had a value. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per liter (mg/L)
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 26 | 29
milligrams per liter (mg/L)
  Cmax | 232 (0.25) | 497 (0.26)
  Ctrough | 78.5 (0.50) | 188 (0.47)

13. Secondary Outcome: AUC(0-inf) and AUC(0-504) After the Sixth Infusion (Week 15, Visit 22)
Description: AUC is defined as the area under the ofatumumab concentration-time curve as a measure of drug exposure. AUC(0-504) is AUC from the start of infusion to 504 hours after the start of the infusion; AUC(0-inf) is AUC from the start of infusion extrapolated to infinity.
Time Frame: Week 15 (Visit 22)
Population: FAS. Data were provided for the number of participants for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams * hours/liter (mg.h/L)
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 25 | 29
Milligrams * hours/liter (mg.h/L)
  AUC(0-inf), n=20, 28 | 177133 (0.41) | 399676 (0.47)
  AUC(0-504), n=24, 28 | 79500 (0.26) | 168866 (0.33)

14. Secondary Outcome: Half Life (t1/2) of Ofatumumab at the Sixth Infusion (Week 15, Visit 22)
Description: Half life is defined as the period of time required for the amount of drug in the body to be reduced by half.
Time Frame: Week 15 (Visit 22)
Population: FAS. Data were provided for the number of participants attending each visit for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 23 | 29
hours | 652 (0.57) | 644 (0.32)

15. Secondary Outcome: CL After the Sixth Infusion (Week 15, Visit 22)
Description: CL is the clearance of drug from plasma, which is defined as the volume of plasma from which the drug is cleared per unit time.
Time Frame: Week 15 (Visit 22)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per hour (mL/h)
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 26 | 29
Milliliters per hour (mL/h) | 6.29 (0.26) | 5.92 (0.33)

16. Secondary Outcome: Vss at the Sixth Infusion (Week 15, Visit 22)
Description: Vss is defined as the volume of distribution at steady state of ofatumumab.
Time Frame: Week 15 (Visit 22)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP
Number analyzed (Participants) | 23 | 29
Liters | 5.15 (0.34) | 5.32 (0.38)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) were collected from the start of study medication until Follow-up (up to 24 months after last treatment). Serious AEs were collected from the start of study medication until study completion (up to 60 months).
Groups:
- 500 mg Ofatumumab + CHOP: Extended Follow-up: Ofatumumab was given on Day 1 and CHOP on Day 3 of each 21-day cycle, with 300 mg in Cycle 1 and 500 mg in Cycles 2 to 6. Participants were followed up for 15 weeks during the Treatment period; then every 3 months for 24 months in the Follow-up period; then every 6 months until Month 60 or withdrawal from the study.
- 1000 mg Ofatumumab + CHOP: Extended Follow-up: Ofatumumab was given on Day 1 and CHOP on Day 3 of each 21-day cycle, with 300 mg in Cycle 1 and 1000 mg in Cycles 2 to 6. Participants were followed up for 15 weeks during the Treatment period; then every 3 months for 24 months in the Follow-up period; then every 6 months until Month 60 or withdrawal from the study.
Arm/Group | 500 mg Ofatumumab + CHOP | 1000 mg Ofatumumab + CHOP | 500 mg Ofatumumab + CHOP: Extended Follow-up | 1000 mg Ofatumumab + CHOP: Extended Follow-up
Serious Adverse Events (participants affected / at risk) | 13/29 | 11/29 | 1/29 | 6/29
Other Adverse Events (participants affected / at risk) | 29/29 | 28/29 | 0/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500 mg Ofatumumab + CHOP (N=29) | 1000 mg Ofatumumab + CHOP (N=29) | 500 mg Ofatumumab + CHOP: Extended Follow-up (N=29) | 1000 mg Ofatumumab + CHOP: Extended Follow-up (N=29)
Leukopenia (Blood and lymphatic system disorders) | 5 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Injection site extravasation (General disorders) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Iliostomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Abnorminal hernia (General disorders) | 0 | 0 | 0 | 2
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Infarction (CNS) (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 500 mg Ofatumumab + CHOP (N=29) | 1000 mg Ofatumumab + CHOP (N=29) | 500 mg Ofatumumab + CHOP: Extended Follow-up (N=29) | 1000 mg Ofatumumab + CHOP: Extended Follow-up (N=29)
Fatigue (General disorders) | 13 | 13 | 0 | 0
Infusion related reaction (General disorders) | 7 | 8 | 0 | 0
Pyrexia (General disorders) | 7 | 8 | 0 | 0
Oedema peripheral (General disorders) | 7 | 6 | 0 | 0
Oedema (General disorders) | 3 | 5 | 0 | 0
Chills (General disorders) | 3 | 3 | 0 | 0
Pain (General disorders) | 2 | 3 | 0 | 0
Asthenia (General disorders) | 2 | 3 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 13 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 12 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 10 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 11 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 11 | 9 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 8 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Polyneuropathy (Nervous system disorders) | 8 | 8 | 0 | 0
Headache (Nervous system disorders) | 6 | 7 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 8 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 6 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 3 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 4 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 7 | 0 | 0
Cystitis (Infections and infestations) | 3 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 10 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 9 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 9 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 1 | 6 | 0 | 0
Hot flush (Vascular disorders) | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 2 | 0 | 0
Hematoma (Vascular disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 0 | 0
Depression (Psychiatric disorders) | 2 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 3 | 2 | 0 | 0
Keratoconjuntivitis sicca (Eye disorders) | 2 | 1 | 0 | 0
Ocular surface disease (Eye disorders) | 0 | 3 | 0 | 0
Eye irritation (Eye disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 3 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Inconsistence (Renal and urinary disorders) | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 2 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.